CLINICAL TRIAL: NCT02940522
Title: A Multi-Center, Randomized, Open-Label Study Comparing Bioavailability When Preservative-free Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) is Administered as an Intramuscular Manual Injection or as a Subcutaneous Injection Using an Auto-injector in Healthy Post-menopausal Women
Brief Title: Comparing Bioavailability When Preservative-free Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL) is Administered as an Intramuscular Manual Injection or as a Subcutaneous Injection Using an Auto-injector in Healthy Post-menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-HPC-PK-010
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Comparing Bioavailability When Makena® is Administered in Healthy Post-menopausal Women
MeSH Terms: interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Subcutaneous (SQ) injection using an autoinjector
  Interventions: Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
- Treatment B (Active Comparator): Intramuscular injection (IM) using syringe and needle
  Interventions: Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)

INTERVENTIONS:
Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
  Other Names: Makena SQ
  Arms: Treatment A
Drug: Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
  Other Names: Makena
  Arms: Treatment B

SUMMARY:
To demonstrate that a single dose of Makena® delivered SQ via auto-injector has comparable bioavailability to a single IM injection of Makena®.

ELIGIBILITY:
Inclusion Criteria:

1. Naturally or surgically postmenopausal women, with or without an intact uterus, aged 50 to 75 years of age, inclusive. FSH levels greater than 40 mIU/mL

Exclusion Criteria:

1. Currently taking any estrogen/progesterone hormone replacement therapy (HRT).
2. History of allergy or sensitivity to hydroxyprogesterone caproate, castor oil or any of the constituents of the study medications, or history of any drug hypersensitivity or intolerance
3. Poorly controlled diabetes.
4. History or current evidence of deep vein thrombosis, pulmonary embolism or arterial thromboembolic disease (e.g., stroke, myocardial infarction).
5. Known, suspected, or current history of carcinoma of the breast.
6. Subjects with a past history of breast cancer on aromatase inhibitors or selective estrogen receptor modulators.
7. Known, suspected, or current history of hormone dependent tumor within the last 5 years.
8. Any current or recent (within previous 12 months) genital bleeding of unknown etiology.
9. Receipt of any investigational drug within 30 days.
10. Receipt of any prescription or OTC medications that are known to alter CYP3A4 or CYP3A5 levels (e.g., carbamazepine, St. John's Wort, ketoconazole, rifampin, ritonavir, alprazolam, azithromycin, loratadine, etc.) within 14.
11. Any estrogen, progestin, or selective estrogen receptor modulator (SERM) treatment within specified time windows before the study start, ranging from 2 to 6 months.
12. High blood pressure at the screening evaluation, defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg.
13. History of excessive alcohol consumption (on average more than 14 units of alcohol/week) during the past 12 months.
14. Use of tobacco products within 30 days of the start of the study.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Krop, MD, Study Chair — AMAG Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Anaheim, California
  - DeLand, Florida
  - Miami, Florida
  - Orlando, Florida
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krop J, Kramer WG. Comparative Bioavailability of Hydroxyprogesterone Caproate Administered via Intramuscular Injection or Subcutaneous Autoinjector in Healthy Postmenopausal Women: A Randomized, Parallel Group, Open-label Study. Clin Ther. 2017 Dec;39(12):2345-2354. doi: 10.1016/j.clinthera.2017.10.020. Epub 2017 Nov 27. PMID 29191450

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: Subcutaneous (SQ) injection using an autoinjector
  Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
- Treatment B: Intramuscular injection (IM) using syringe and needle
  Makena® (Hydroxyprogesterone Caproate Injection, 250 mg/mL)
Period: Overall Study
Arm/Group | Treatment A | Treatment B
Started | 59 | 61
Completed | 57 | 59
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 53 | 100
  >=65 years | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.16) | 57.0 (5.68) | 58.4 (6.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 61 | 120
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Areas Under the Curve (AUC) to the Last Time With a Concentration ≥ LLOQ [AUC0-t] and to Infinity [AUCinf]
Description: Comparison of areas under the curve (AUC) to the last time with a concentration ≥ LLOQ [AUC0-t] and to infinity [AUCinf] for the Primary PK Population
Time Frame: 9 weeks
Population: The Primary PK Population consisted of 45 subjects each for both treatments for whom whole blood was analyzed. Subjects were excluded from Treatment A and Treatment B due to insufficient number of samples for planned analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr x ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 45 | 45
hr x ng/mL
  AUC(0-t) | 2,313 (23.5) | 2,098 (27.7)
  AUC(inf): number analyzed (Participants) | 39 | 41
  AUC(inf) | 2,469 (22.8) | 2,175 (27.8)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Comparison of bioavailability; The PK parameters were compared between treatments using an analysis of variance statistical model with treatment as the fixed effect, using the natural logarithms of the data. As the objective was to assess whether comparable exposure could be obtained using the higher SQ dose, the data were not normalized for dose before the statistical analysis

2. Primary Outcome: Comparison of the Maximum Plasma Concentration (Cmax)
Description: Comparison of the maximum plasma concentration (Cmax) for the Primary PK Population
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 45 | 45
ng/mL | 7.88 (71.9) | 6.91 (62.9)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Comparison of bioavailability data; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Comparison of Tmax
Description: Comparison of PK parameter Tmax for the Primary PK population
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: hr
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 45 | 45
hr | 48.1 [18 to 342] | 49.7 [2 to 336]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Comparison of bioavailability data; [other analysis details as in outcome 1, analysis 1]

4. Secondary Outcome: Comparison of AUC (0-168)
Description: Comparison of PK Parameter AUC (0-168) for the Primary PK Population
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr x ng/mL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 45 | 45
hr x ng/mL | 813 (41.5) | 790 (55.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Comparison of bioavailability data; [other analysis details as in outcome 1, analysis 1]

5. Secondary Outcome: Comparison of t1/2
Description: Comparison of PK parameter t1/2 for the Primary PK Population
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 39 | 41
hr | 212 (29.1) | 185 (25.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Comparison of bioavailability data; [other analysis details as in outcome 1, analysis 1]

6. Secondary Outcome: Comparison of Elimination Rate Constant
Description: Comparison of the elimination rate constant for the Primary PK Population
Time Frame: 9 weeks
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 39 | 41
1/hr | 0.0033 (29.1) | 0.0038 (25.5)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Other — Comparison of bioavailability data; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 9 weeks.
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/61
Other Adverse Events (participants affected / at risk) | 32/59 | 23/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=59) | Treatment B (N=61)
Injection site pain (General disorders) | 22 (25) | 5 (6)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site discoloration (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Injection site paraesthesia (General disorders) | 1 (1) | 0 (0)
Injection site pruritis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vessel puncture site reaction (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (9) | 10 (10)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No